CLINICAL TRIAL: NCT00001979
Title: Studies of Immunologically-Mediated Kidney Diseases
Brief Title: Immune System Related Kidney Disease
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920156; 92-DK-0156
Record Dates: First submitted 2000-01-20; First posted 2000-01-21 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-05-15

CONDITIONS: Kidney Disease; Nephrotic Syndrome
Keywords: Kidney Disease; Chronic Kidney Disease; Natural History
MeSH Terms: conditions — Kidney Diseases; Nephrotic Syndrome; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with known or suspected immunologically-mediated kidney diseases or immunologically-mediated diseases with potential for kidney disease.

SUMMARY:
Kidney diseases related to the immune system include, nephrotic syndrome, glomerulonephritis, membranous nephropathy, lupus nephritis, and nephritis associated with connective tissue disorders.

This study will allow researchers to admit and follow patients suffering from autoimmune diseases of the kidney. It will attempt to provide information about the causes and specific abnormalities associated with autoimmune kidney disease.

Patients with kidney disease as a result of their immune system, and patients with diseases of the immune system who may later develop kidney disease, will be potential subjects for this study.

Patients will undergo a history and physical examination, and standard laboratory test to more closely understand the causes, signs, symptoms, and responses to medication of these diseases. Based on these evaluations the patients may qualify as candidates for other experimental studies. At any time these patients may be asked to submit blood or urine samples for further research.

DETAILED DESCRIPTION:
Study Description:

This study evaluates participants with known or suspected immunologically-mediated kidney diseases, including but not limited to nephrotic syndrome, glomerulonephritis, membranous nephropathy, lupus nephritis, and nephritis associated with other systemic or connective tissue disorders. Participants who have immunologically-mediated diseases with potential for kidney disease will be evaluated as well. Studies will include characterization of the clinical and laboratory features of these disorders, studies of natural history and complications, evaluation of responses to standard treatment. Blood and urine samples will be collected for immunological research conducted under this protocol.

Objectives:

Primary:

-To collect samples and data obtained during standard clinical care that can be used to better understand rare forms of immunologically-mediated renal disorders, atypical renal disease that have not been fully characterized, and to allow for future research studies.

Exploratory:

* Characterize immunologically-mediated kidney diseases with regard to immune dysregulation, immune cell populations and role of complement activation.
* Development of assays for novel antibodies.
* Search for additional antibodies involved in the pathogenesis of membranous nephropathy and other glomerular diseases.
* Assess changes in metabolic (e.g. vitamin D, lipids) and endocrine function (e.g. thyroid, adrenal function) during the evolution of the nephrotic state, during treatment and during remission.
* Identify disease-causing memory B cells in participants with membranous nephropathy and correlation with membranous nephropathy relapse. Assess biological effects of phospholipase A2-receptor antibody epitope on the isolated memory B-cells.
* Compare immune cell types, including B and T cell populations and cell type specific markers in the pathogenesis of immune-mediated kidney disease.
* Compare changes in metabolome and proteome of urine and blood during the nephrotic syndrome, during treatment and in remission.
* Computational analysis of renal structures which may provide predictive methods that would discriminate progressors from non-progressors beyond sclerosis in membranous nephropathy.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, a participant must meet all of the following criteria:

1. Adults >= 18 years of age and children 10-17 years of age
2. Participants with

   1. known, proven, or suspected immunologically-mediated kidney diseases, including but not limited to nephrotic syndrome, glomerulonephritis, membranous nephropathy, lupus nephritis, and nephritis associated with other systemic or connective tissue disorders, OR
   2. immunologically-mediated diseases with the potential for kidney disease.
3. Ability of the participant or guardian to understand and the willingness of the participant or guardian to provide written informed consent.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Concomitant medical problems which would confound the interpretation of studies of the immunologic kidney disorder.
2. Concomitant medical, surgical, or other conditions for which inadequate facilities or funds are available to support their care at the NIH.

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with known or suspected immunologically-mediated kidney diseases, including but not limited to, nephrotic syndrome, glomerulonephritis, membranous nephropathy, lupus nephritis, and nephritis associated with other systemic or connective tissue disorders, or immunologically-mediated diseases with the potential for kidney disease.@@@
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1992-06-25 (Actual)

PRIMARY OUTCOMES:
Provision of biospecimens | ongoing
  Patients with autoimmune diseases for whom there are no current experimental treatment protocols can be admitted for study and follow-up; they will provide a ready pool of candidates who can be asked to provide blood specimens for ongoing laboratory studies.

CONTACTS AND LOCATIONS:
Overall Officials: Meryl A Waldman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1992-DK-0156.html